CLINICAL TRIAL: NCT02111408
Title: Stroke - Sleep Disorders, Dysfunction of the Autonomic Nervous System and Depression
Status: Completed | Type: Observational
Sponsor: Helle Klingenberg Iversen, MD, DmSc (Other)
Responsible Party: Sponsor-Investigator, Helle Klingenberg Iversen, MD, DmSc, M.D., Glostrup University Hospital, Copenhagen
Organization: Glostrup University Hospital, Copenhagen (Other)
Other Study IDs: VEK: H-2-3013-091; H-2-3013-091 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-04-03; First posted 2014-04-11 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Sleep apnea syndromes; Autonomic nervous system +/- disease; Depression; Peripheral arterial disease
MeSH Terms: conditions — Stroke; Sleep Apnea Syndromes; Depression; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute stroke: No interventions. Only tests for depression, sleepapnea and autonomic dysfunction.

SUMMARY:
The purpose of this study is to investigate sleep disordered breathing, autonomic dysfunction, and post stroke depression in acute and chronic stroke patients. Furthermore, to explore the interaction between these comorbidities, and their relation to stroke aetiology.

DETAILED DESCRIPTION:
Up to fifty percent of stroke patients suffer less noticeable comorbidities after the acute phase of a stroke and often the rest of their life. It concerns sleep disordered breathing (SDB), post stroke depression (PSD), and dysfunction of the autonomic nervous system. These comorbidities are seldom recognized, but are associated with a poorer outcome after stroke, reduced quality of life as well as an increased risk of new vascular events.

Little is known about the course of the comorbidities, the relationship between the mentioned diseases or which patients are more commonly affected.

The investigators will investigate the following hypotheses, and assess the results compared to the stroke aetiology:

1. Stroke patients with SDB have an impaired autonomic function
2. Stroke patients with SDB have an increased risk of PSD
3. Stroke patients with autonomic dysfunction have an increased risk of PSD

The investigators will examine stroke patients for signs of sleep disordered breathing, autonomic dysfunction and depression, both in the acute phase (days), in the chronic phase (months) and the very chronic state (years). Thereby the investigators can map the comorbidities course over time. At the same time the patients will be tested for peripheral small and large artery disease as well as MRI will be used to investigate sign of cerebral small vessel disease.

Based on power calculations 335 individuals will be enrolled in order to satisfy the project requirements.

ELIGIBILITY:
Inclusion Criteria:

• Clinical stroke either ischaemic or haemorrhagic

Exclusion Criteria:

* Transitory ischemic attac
* Congenital or acquired brain disease, other than stroke
* Dementia
* Mental retardation
* Fatal stroke or severe comorbidities with short expected life
* Pregnancy or breastfeeding
* Altered consciousness e.g. delirium or status epilepticus
* Other cause of the patient, according to the investigator believes, can not complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is recruited among patients admitted at the acute stroke unit at Glostrup university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-03; Primary Completion 2017-02 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Sleep disordered breathing at any time after stroke. | six month after stroke
  The test for sleep disordered breathing will be performed within 7 days from stroke onset and after 6 month and five years.
  Mild sleep apnea if AHI between 5 and 15, moderate sleep apnea if AHI between 15 and 30 and severe sleep apnea if AHI above 30. Subdivided into obstructive, central or mixed.
Autonomic dysfunction at any time after stroke. | six month after the stroke
  The test for autonomic dysfunction will be performed within 7 days from stroke onset and after 6 month and five years.
  Abnormal result of the valsalva manoeuvre, deep breathing, active standing or tilt table test. Improvement or worsening of the parameters like HRV, BRS and CO during the study period.
Depression at any time after stroke | six month after the stroke
  The test for depression will be performed within 7 days from stroke onset and after 6 month and five years.
  Mild, moderate or severe depression according to HAM-D6, MDI or HADS

SECONDARY OUTCOMES:
Peripheral artery disease at any time after stroke | six month after the stroke
  The tests will be performed within 7 days from stroke onset and after 6 month and five years.
  Stenosis of the carotid artery, abnormal ankle-brachial index or endothelial dysfunction.

OTHER OUTCOMES:
New vascular episodes at any time after stroke | Assessed at follow-up after six month
  Assessed at follow-up after six month and five years. Stroke, TIA, acute coronary syndrome or operation for peripheral vascular disease.
Death by cause at any time after stroke | Assessed at follow-up after six month
  Assessed at follow-up after six month and five years

CONTACTS AND LOCATIONS:
Overall Officials: Helle Iversen, MD, DMSc, Principal Investigator — Stroke research, Glostrup hospital
Locations (1):
- Department of clinical stroke research, department of neurology, Glostrup Hospital, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simonsen SA, Andersen AV, West AS, Wolfram F, Jennum P, Iversen HK. Sleep-disordered breathing and cerebral small vessel disease-acute and 6 months after ischemic stroke. Sleep Breath. 2022 Sep;26(3):1107-1113. doi: 10.1007/s11325-021-02482-1. Epub 2021 Sep 2. PMID 34476728